CLINICAL TRIAL: NCT00294593
Title: One-year Double-blind Placebo-controlled Phase 2-3 Study to Evaluate the Effect of Oral Folinic Acid Treatment (1mg/kg/d) on the Psychomotor Development of Young Down Syndrome Patients
Brief Title: Efficacy Study of Folinic Acid to Improve Mental Development of Children With Down Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut Jerome Lejeune (Other)
Collaborators: Fondation Jérôme Lejeune (Other)
Responsible Party: Franck Sturtz, Institut Jerome Lejeune
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IJL-FA-TH01
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Down Syndrome
Keywords: Down syndrome; folinic acid therapy; cognitive functions
MeSH Terms: conditions — Down Syndrome | interventions — Leucovorin

INTERVENTIONS:
Drug: folinic acid

SUMMARY:
The purpose of this study is to determine whether folinic acid can improve developmental quotient of young Down syndrome patients, given that these present signs of folate deficiency which are known to cause reversible neurological, psychiatric and cognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome without mosaicism
* age 3 to 30 months
* weight over 4 kg
* possible assessment by the revised Brunet-Lezine scale

Exclusion Criteria:

* history of leukemia
* West syndrome or non-stable epilepsy
* non-stable thyroxin treatment

Ages: 3 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120
Dates: Start 2000-10; Study Completion 2003-12

PRIMARY OUTCOMES:
Score on a psychomotor development scale after a 6 and 12 months treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henri Blehaut, M.D., Study Director — Institut Jerome Lejeune; Clotilde Mircher, MD, Principal Investigator — Institut Jerome Lejeune
Locations (1):
- Institut Jerome Lejeune, Paris, France

REFERENCES:
- [Background] Botez MI, Botez T, Leveille J, Bielmann P, Cadotte M. Neuropsychological correlates of folic acid deficiency: facts and hypotheses. In: Botez MI, Reynolds EH, eds. Folic acid in neurology, psychiatry and internal medicine. New York, Raven Press, 1979:435-461.
- [Background] Lejeune J. [Pathogenesis of mental impairment in trisomy 21]. Ann Genet. 1991;34(2):55-64. French. PMID 1836122
- [Derived] Blehaut H, Mircher C, Ravel A, Conte M, de Portzamparc V, Poret G, de Kermadec FH, Rethore MO, Sturtz FG. Effect of leucovorin (folinic acid) on the developmental quotient of children with Down's syndrome (trisomy 21) and influence of thyroid status. PLoS One. 2010 Jan 11;5(1):e8394. doi: 10.1371/journal.pone.0008394. PMID 20084109